CLINICAL TRIAL: NCT01583699
Title: Confocal Laser Endomicroscopy as Diagnostic Tool for Gastrointestinal MALT-lymphoma
Brief Title: Endomicroscopy and Gastric MALT-lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Werner Dolak, MD, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EK 111/2011
Record Dates: First submitted 2012-01-08; First posted 2012-04-24 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: MALT-lymphoma
Keywords: MALT-lymphoma; Confocal laser endomicroscopy; Gastrointestinal endoscopy
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endomicroscopy (Experimental): All patients included into the study will undergo endomicroscopy of the upper GI-tract.
  Interventions: Procedure: Confocal laser endomicroscopy; Device: Confocal Laser Endomicroscope

INTERVENTIONS:
Procedure: Confocal laser endomicroscopy — Endomicroscopy of the upper gastrointestinal tract to capture endomicroscopic pictures from the small bowel, stomach and esophagus.
Device: Confocal Laser Endomicroscope — Pentax EC-3870 CIFK with the ISC-1000 confocal endomicroscopy processor - Pentax, Tokyo, Japan and Optiscan Pty Ltd, Notting Hill, Victoria, Australia

SUMMARY:
Extranodal marginal zone B-cell lymphoma (MZBL) of the mucosa associated lymphoid tissue (MALT-lymphoma) represents a distinct clinical entity and is the most common form of extranodal lymphoma, with a predilection for the stomach. About 90% of gastric MALT-lymphomas are associated with infection with Helicobacter pylori (HP) and eradication of the pathogen leads to regression of the tumor in a high percentage of patients at early tumour stages. Nevertheless, following complete remission after HP-eradication, the risk of relapse justifies lifelong follow-up examinations. Supported by recent findings at the investigators department, endoscopic controls should include a close examination of the small bowel, as relapses can involve different gastrointestinal sites. To continue the investigators diagnostic approach as well as to further improve the detection rate of MALT-lymphoma relapses, the investigators plan to introduce the novel confocal laser endomicroscope (CLE) into the diagnostic management of MALT-lymphoma patients. In the context of a prospective clinical pilot trial the investigators aim to establish MALT-lymphoma specific CLE-markers that can be used for the in vivo diagnosis of the disease. Comparing endomicroscopic findings, drawn from the stomach and small bowel of 50 MALT-lymphoma patients who will undergo staging or follow up endoscopies at the investigators department, to the histological evaluation of biopsy samples as present gold standard, the investigators want to determine whether CLE can provide reliable data for the accurate detection of MALT-lymphoma associated changes. Endomicroscopic aspects of patients with chronic gastritis, gastric adenocarcinoma and healthy subjects should serve as controls. In comparison to random biopsies which represent the current standard, the investigators aim to prove, whether endomicroscopy will find MALT-lymphoma lesions more accurately and thus help to spare patients unnecessary biopsies.

DETAILED DESCRIPTION:
Introduction

Extranodal marginal zone B-cell lymphoma (MZBL) of the mucosa associated lymphoid tissue (MALT-lymphoma) is the most common form of extranodal lymphoma [1, 2]. Although MALT-lymphoma may involve different organs, the stomach represents the site of predilection of this malignant disease. About 90% of gastric MALT-lymphomas are associated with infection with Helicobacter pylori (HP) [3] and eradication of the pathogen leads to tumor regression in a high percentage of patients at early tumor stages [4, 5]. Relapses after HP-eradication and primary advanced tumor stages require chemotherapeutic treatment, radiation therapy and, in some cases, surgery [6]. Following complete remission lifelong follow-up examinations should be performed in order to detect relapses [7].

Histologically, MALT-lymphoma is characterized by an infiltration of the lamina propria by lymphomatous centrocyte-like cells that spread into the surrounding mucosal layers [8]. In immunohistochemistry they show CD 20 positive staining properties. When they spread to lymph nodes or spleen they accumulate typically within the marginal zone (for this reason they are classified as "marginal zone lymphoma") [2]. Dissemination to other organs, especially to other mucosal sites may occur frequently wherefore detailed diagnostics are required during MALT-lymphoma staging and follow-up. Spreading within the gastrointestinal tract (GI-tract), to the small bowel, for example, is rare, but can be assessed very easily with standard endoscopic procedures as recently reported at our department [9].

For gastric MALT-lymphoma gastroscopy with biopsy assessment is the current follow-up examination of choice. Multiple biopsies should be taken randomly from all gastric sites and specifically from all suspicious lesions. Recent developments for the enhancement of the tissue contrast during the endoscopic examinations (chromoendoscopy or Narrow Band Imaging, for example) helped to detect MALT-lymphoma lesions. Nevertheless, detection rates hardly changed, since all these techniques rely on the presence of superficial features[10].

An endoscopic technique that allows an evaluation of deeper wall layers is endoscopic ultrasonography. During the last years it has become an important amending tool in the diagnostic management of gastric MALT-lymphoma. Although it provides essential information about tumor infiltration depth and lymph node involvement in the context of staging procedures, it cannot replace histological assessment during follow-up, since endosonographic findings do not show a good correlation to histological results over time [11, 12].

The newest development that has been introduced in the endoscopic management of the gastrointestinal tract is the so called confocal laser endomicroscope (CLE). Confocal microscopy was developed by Marvin Minsky in the late 1950s. Its principle is the microscopic scanning of focal points below the surface of an object. In comparison to conventional light microscopy it uses a special filter system to avoid image overlapping by surrounding tissue. In detail, a light source (normally a laser) is focused by a microscope objective lens to a diffraction limited spot on or inside the object. Light that is scattered, or fluorescence excited (achieved through fluorescein staining, for example) and emitted, at the focus in the sample will partially return back through the optics along the path from which it arrived. A beam-splitter placed into the path reflects the return light towards a detector. The optics will focus the light from the focal point in the specimen to its conjugate focus near the detector (hence the technology is termed "con-focal"). Here a spatial filter ("pinhole") is used to extinguish all light deriving from areas outside the focal point. Light reflections from the focal point itself will be forwarded to the detector which is connected to a computer system that digitalises the optical signal and creates the in vivo histological image [13].

Focusing on its clinical impact, confocal microscopy is the first technique to allow in vivo evaluation of tissue structures beneath their surface. Because of many breakthroughs in miniaturisation (mostly in the 1990s) this technology could be applied for intraluminal use in gastroenterology, integrated into an otherwise standard endoscope. It allows the in vivo histological visualisation of the upper 250 micrometers of all walls within the gastrointestinal tract, additionally to the normal function of white light endoscopy (provided by two separate screens on top of the workstation) [13].

The in vivo visualisation of different GI-pathologies led to the first publications on the clinical use of CLE. Kiesslich et al., as one of the pioneers of the technique, published a case on live imaging of Helicobacter pylori by CLE in the stomach [14]. At our department we recently reported the endomicroscopic findings of a patient with Whipple's disease. Detecting foamy macrophages within the lamina propria which were clearly distinguishable from goblet cells in the surrounding CLE could provide in vivo histology at the single cell level [15].

Assessing GI-pathologies more systematically there have been many publications dealing with the use of CLE in the context of follow-up examinations of conditions that predispose to the development of malignancies. For Barrett's oesophagus, for example, Kiesslich et al. found high sensitivity and specificity rates for the detection of Barrett's metaplasia as well as for the prediction of Barrett's associated neoplastic changes - for both results CLE derived pictures were compared to conventional histology [16]. In a first prospective, randomized, double-blind, controlled, crossover trial Dunbar et al. proved these findings, as CLE-targeted biopsies had a higher diagnostic yield for Barrett's oesophagus associated neoplasia than standard endoscopy with 4-quadrant random biopsy [17]. Similar results have already been published for patients with ulcerative colitis that were routinely screened for colon cancer. It could be shown that CLE is a useful tool to improve the diagnostic yield. At the same time, it helped to take conventional biopsies more accurately, which can spare patients unnecessary biopsies [18].

Combining the potential of CLE to improve the diagnostic yield during surveillance with its properties of scanning the upper 250µm of the GI-wall (which equates nearly the whole depth of the mucosa) makes it the ideal tool for the diagnostic management of gastric MALT-lymphoma, where pathologies typically arise from the lamina propria, a deeper layer of the mucosa [8].

Study Aims

In this clinical pilot study the investigators aim to examine patients with gastric MALT-lymphoma by confocal laser endomicroscopy (CLE) in the context of staging or follow-up endoscopies. To our knowledge no systematic study on the use of CLE in MALT-lymphoma patients has yet been performed.

* The investigators aim to determine whether the diagnosis of MALT-lymphoma can be achieved by evaluating endomicroscopic features of suspicious lesions of both the stomach and the small bowel, as these GI-parts are easily accessible by upper endoscopy. Conventional biopsies from the GI-parts observed should serve as comparable gold standard.
* Including endomicroscopic results of patients with chronic gastritis, gastric adenocarcinoma and healthy subjects as controls the investigators aim to establish MALT-lymphoma specific markers that can be used for a "biopsy-free" in vivo diagnosis of the disease.

Study Design

Prospective clinical trial without randomisation or blinding

Study Population

Patients referred to our department for upper endoscopy in the context of staging or follow-up of gastric MALT-lymphoma.

Exclusion criteria:

* patients allergic to one of the drug components (including drugs used for conscious sedation like propofol or midazolam as well as fluorescein, the fluorescent dye used for CLE )
* refusal to participate in the study
* patient's age below 18 years

Methods

This investigation will be performed at the Division of Gastroenterology and Hepatology, Department of Internal Medicine III., in close cooperation with the Division of Oncology, Department of Internal Medicine I. and the Clinical Institute of Pathology at the Medical University of Vienna.

As this study has been planned as a pilot trial, it mainly focuses on the qualitative endomicroscopic features drawn from our examinations to yield reference pathologies for accurate diagnosis in the future. Nevertheless, a quantitative analysis will be performed by comparing CLE-derived diagnoses with histological results to calculate sensitivity and specificity of CLE based MALT-lymphoma diagnosis. Based on current incidence and relapse rates of the disease the investigators estimated to include 50 patients in order to get a meaningful patient sample for qualitative and quantitative analysis. Given the current number of MALT-lymphoma patients who undergo staging or follow-up endoscopies at the investigational site, this patient sample can be included within a period of two years.

All patients who fulfill the listed inclusion criteria, will receive the patient information form of this study together with the usual informed consent form of the respective endoscopic examination they are about to undergo. Patient information will be done at least 24 hours before the intervention, as practised at our unit. If the patient agrees to participate in the study he will be prepared for endoscopy with our confocal laser endomicroscope (Pentax EC3870K with the ISC-1000 confocal endomicroscopy processor - Pentax, Tokyo, Japan and Optiscan Pty Ltd, Notting Hill, Victoria, Australia) by administration of intravenous propofol and/or midazolam as routinely used for conscious sedation during endoscopic procedures at our department. Additionally, 5-10 ml of a 10% solution of fluorescein sodium will be administered intravenously to enhance tissue fluorescence during endomicroscopy.

All drugs will be administered by medical specialists, assistant doctors or registered nurses, as routinely practiced at our institution.

CLE picture capturing will start at the deepest point reachable in the small bowel. During withdrawal of the scope CLE pictures will be taken every 10 centimetres in the small bowel, then from the antrum and body of the stomach and from the esophagus. Furthermore, CLE will be applied for distinct looking areas, suspicious of pathologic origin. Wherever CLE pictures are obtained, a conventional biopsy will be taken from the same localisation.

CLE pictures will be captured and stored routinely using our standard data management system. They will be evaluated immediately during the endoscopic procedure together with a board certified GI-pathologist, who will establish an initial diagnosis.

Conventional biopsies will be processed and evaluated according to the criteria as outlined in the recent WHO-classification for MALT-lymphoma. In all patients, immunologic phenotyping on paraffin sections will be done for demonstration of light chain restriction and for the phenotype CD20+CD5-CD10-cyclinD1- which, in context with the microscopic appearance, is consistent with MALT-lymphoma. In addition, all patients will be assessed for MALT-lymphoma specific translocations, especially t(11;18)(q21;q21).

Endomicroscopic controls (patients with chronic gastritis, gastric adenocarcinoma and healthy subjects) will be collected from present data of endomicroscopic procedures already performed within routine examinations.

At the end of the study all CLE pictures and histological cuts will be evaluated separately by two blinded board certified pathologists. In case of discordant diagnoses they will analyse the respective cases together to reach an agreement on the final diagnosis. All cases where the initial and the final diagnosis are deviating from each other will be re-evaluated together by all specialists involved.

Ethical implications

Confocal laser endomicroscopy is a safe new technique that has already been studied in clinical trials [16, 17]. Its safety is being guaranteed by the use of low intensity laser light that can at worst cause local bleaching of fluorescein containing cells, which is harmless, reversible and even used as diagnostic sign in experimental conditions [13].

This study protocol had been already approved by the ethics commission of the Medical University of Vienna. All procedures in the context of this study will be performed in accordance to the Declaration of Helsinki as well as to the guidelines for Good Scientific Practice (GSP) of the Medical University of Vienna.

Expected impact and Outlook

If the investigators find MALT-lymphoma specific markers that can be used for a "biopsy-free" in vivo diagnosis, this could lead to another reduction of invasive procedures for the affected patients which may have an important clinical impact, as biopsy assessment is often limited by the rather bad coagulation status of oncologic patients.

In case the study aims will be supported by the results of this pilot trial, a randomized controlled trial comparing in vivo diagnosis to conventional histological assessment in matters of diagnostic yield will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to our department for upper endoscopy in the context of staging or follow-up of gastric MALT-lymphoma.

Exclusion criteria:

* patients allergic to one of the drug components (including drugs used for conscious sedation like propofol or midazolam as well as fluorescein, the fluorescent dye used for CLE )
* refusal to participate in the study
* patient's age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Qualitative MALT-features on Endomicroscopy | 2 years
  Establishing endomicroscopic features of MALT-lymphoma in the upper gastrointestinal tract. This outcome is a qualitative endpoint that will be assessed only descriptively.

SECONDARY OUTCOMES:
Sensitivity and Specificity of Endomicroscopy to diagnose GI-MALT-Lymphoma | 2 years
  At the end of the study, endomicroscopic pictures gained during the study will be assessed by two blinded pathologists regarding judgement on MALT-lymphoma presence or absence. The results will be compared to the corresponding histological sections in order to calculate sensitivity ans specificity for the technique.

CONTACTS AND LOCATIONS:
Overall Officials: Werner Dolak, MD, Principal Investigator — Medical University of Vienna, Department of Internal Medicine III, Division of Gastroenterologie and Hepatologie; Andreas Puespoek, m, Study Director — Medical University of Vienna, Department of Internal Medicine III, Division of Gastroenterology and Hepatology; Markus Raderer, MD, Study Chair — Medical University of Vienna, Department of Internal Medicine I, Division of Oncology
Locations (1):
- Medical University of Vienna, Department of Internal Medicine III, Division of Gastroenterology and Hepatology, Vienna, Austria

REFERENCES:
- [Background] Ott G, Balague-Ponz O, de Leval L, de Jong D, Hasserjian RP, Elenitoba-Johnson KS. Commentary on the WHO classification of tumors of lymphoid tissues (2008): indolent B cell lymphomas. J Hematop. 2009 Jul;2(2):77-81. doi: 10.1007/s12308-009-0037-9. Epub 2009 Jun 25. PMID 19669189
- [Background] Ferreri AJ, Zucca E. Marginal-zone lymphoma. Crit Rev Oncol Hematol. 2007 Sep;63(3):245-56. doi: 10.1016/j.critrevonc.2007.04.009. Epub 2007 Jun 20. PMID 17583528
- [Background] Morgner A, Schmelz R, Thiede C, Stolte M, Miehlke S. Therapy of gastric mucosa associated lymphoid tissue lymphoma. World J Gastroenterol. 2007 Jul 14;13(26):3554-66. doi: 10.3748/wjg.v13.i26.3554. PMID 17659705
- [Background] Zullo A, Hassan C, Andriani A, Cristofari F, De Francesco V, Ierardi E, Tomao S, Morini S, Vaira D. Eradication therapy for Helicobacter pylori in patients with gastric MALT lymphoma: a pooled data analysis. Am J Gastroenterol. 2009 Aug;104(8):1932-7; quiz 1938. doi: 10.1038/ajg.2009.314. Epub 2009 Jun 16. PMID 19532131
- [Background] Terai S, Iijima K, Kato K, Dairaku N, Suzuki T, Yoshida M, Koike T, Kitagawa Y, Imatani A, Sekine H, Ohara S, Shimosegawa T. Long-term outcomes of gastric mucosa-associated lymphoid tissue lymphomas after Helicobacter pylori eradication therapy. Tohoku J Exp Med. 2008 Jan;214(1):79-87. doi: 10.1620/tjem.214.79. PMID 18212490
- [Background] Raderer M, Isaacson PG. Extranodal lymphoma of MALT-type: perspective at the beginning of the 21st century. Expert Rev Anticancer Ther. 2001 Jun;1(1):53-64. doi: 10.1586/14737140.1.1.53. PMID 12113133
- [Background] Raderer M, Streubel B, Woehrer S, Puespoek A, Jaeger U, Formanek M, Chott A. High relapse rate in patients with MALT lymphoma warrants lifelong follow-up. Clin Cancer Res. 2005 May 1;11(9):3349-52. doi: 10.1158/1078-0432.CCR-04-2282. PMID 15867234
- [Background] Isaacson PG. Gastric MALT lymphoma: from concept to cure. Ann Oncol. 1999 Jun;10(6):637-45. doi: 10.1023/a:1008396618983. PMID 10442184
- [Background] Dolak W, Raderer M, Maresch J, Muellauer L, Puespoek A, Chott A, Haefner M. Detection of gastric MALT lymphoma spreading to the small bowel by enteroscopy. Endoscopy. 2011 Aug;43(8):731-3. doi: 10.1055/s-0030-1256435. Epub 2011 Jun 7. PMID 21656457
- [Background] Hyatt BJ, Paull PE, Wassef W. Gastric oncology: an update. Curr Opin Gastroenterol. 2009 Nov;25(6):570-8. doi: 10.1097/MOG.0b013e328331b5c9. PMID 19816172
- [Background] Puspok A, Raderer M, Chott A, Dragosics B, Gangl A, Schofl R. Endoscopic ultrasound in the follow up and response assessment of patients with primary gastric lymphoma. Gut. 2002 Nov;51(5):691-4. doi: 10.1136/gut.51.5.691. PMID 12377808
- [Background] Al-Taie OH, Dietrich CF, Dietrich CG, Fischbach W. [Role of endoscopic ultrasound in gastrointestinal lymphomas]. Z Gastroenterol. 2008 Jun;46(6):618-24. doi: 10.1055/s-2008-1027517. German. PMID 18537089
- [Background] Kiesslich R, Galle P, Neurath M. Atlas of endomicroscopy. Springer Medical Publishing. 2008
- [Background] Kiesslich R, Goetz M, Burg J, Stolte M, Siegel E, Maeurer MJ, Thomas S, Strand D, Galle PR, Neurath MF. Diagnosing Helicobacter pylori in vivo by confocal laser endoscopy. Gastroenterology. 2005 Jun;128(7):2119-23. doi: 10.1053/j.gastro.2004.12.035. PMID 15940642
- [Background] Dolak W, Leitner J, Maresch J, Wrba F, Mueller C. In vivo identification by confocal laser endoscopy of foamy macrophages associated with Whipple's disease. Endoscopy. 2010;42 Suppl 2:E310-1. doi: 10.1055/s-0030-1255809. Epub 2010 Nov 26. No abstract available. PMID 21113886
- [Background] Kiesslich R, Gossner L, Goetz M, Dahlmann A, Vieth M, Stolte M, Hoffman A, Jung M, Nafe B, Galle PR, Neurath MF. In vivo histology of Barrett's esophagus and associated neoplasia by confocal laser endomicroscopy. Clin Gastroenterol Hepatol. 2006 Aug;4(8):979-87. doi: 10.1016/j.cgh.2006.05.010. Epub 2006 Jul 13. PMID 16843068
- [Background] Dunbar KB, Okolo P 3rd, Montgomery E, Canto MI. Confocal laser endomicroscopy in Barrett's esophagus and endoscopically inapparent Barrett's neoplasia: a prospective, randomized, double-blind, controlled, crossover trial. Gastrointest Endosc. 2009 Oct;70(4):645-54. doi: 10.1016/j.gie.2009.02.009. Epub 2009 Jun 25. PMID 19559419
- [Background] Kiesslich R, Goetz M, Lammersdorf K, Schneider C, Burg J, Stolte M, Vieth M, Nafe B, Galle PR, Neurath MF. Chromoscopy-guided endomicroscopy increases the diagnostic yield of intraepithelial neoplasia in ulcerative colitis. Gastroenterology. 2007 Mar;132(3):874-82. doi: 10.1053/j.gastro.2007.01.048. Epub 2007 Jan 31. PMID 17383417
- [Derived] Dolak W, Kiesewetter B, Mullauer L, Mayerhoefer M, Troch M, Trauner M, Hafner M, Raderer M, Puspok A. A pilot study of confocal laser endomicroscopy for diagnosing gastrointestinal mucosa-associated lymphoid tissue (MALT) lymphoma. Surg Endosc. 2016 Jul;30(7):2879-85. doi: 10.1007/s00464-015-4572-4. Epub 2015 Oct 20. PMID 26487230